CLINICAL TRIAL: NCT01467960
Title: Detection of Apolipoprotein D (ApoD) in Human Serum as Marker of Parkinson's Disease
Brief Title: Apolipoprotein D (ApoD) In Human Serum As Marker Of Parkinson's Disease
Acronym: ApoD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Privatklinik Villa Melitta (Other)
Responsible Party: Principal Investigator, Andreas Waldner, Study Director, Privatklinik Villa Melitta
Other Study IDs: Melitta-ApoD-2011
Record Dates: First submitted 2011-10-30; First posted 2011-11-09 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson's
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Group I: Healthy Subjects aged 20-40
- Group II: Healthy Subjects aged 40-65
- Group III: Healthy Subjects aged more than 65
- Group A: Patients at Stage I, H&Y classification
- Group B: Patients at Stage II, H&Y classification
- Group C: Patients at Stage more than III, H&Y classification

SUMMARY:
In Italy affected people are 200,000 and every year Parkinson new cases are 10,000. Aging is the principle risk factor of Parkinson with the possibility of its development doubling every five years after 65. Because of the increase of the social longevity and aging as the main risk factor, there are many repercussions on the health system (hospital stays and pharmaceutical costs) as on the social system (assistance- related problems). Parkinson's disease exerts an extremely negative impact on life's quality of the patient. In fact, because of Parkinson symptoms (tremor, dribble, etc), patient's social life will be reduced with the consequent development of the depression. Consequently, the early detection and treatment of Parkinson's is necessary.

To achieve this goal, Apolipoprotein D (ApoD) in human serum as a marker of the oxidative stress-inflammation vicious cycle seems most promising candidate for diagnosis.

DETAILED DESCRIPTION:
Total participants: n=180.

Study Part 1:

Health persons: n=90; Groups of health persons: n=3; Subjects per group: n=30.

Study Part 2:

Patients: n=90; Groups of patients: n=3; Subjects per group: n=30.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease in the pathological related stages (Hoehn and Yahr)
* Persons > 20 years

Exclusion Criteria:

* Patients with a neurodegenerative disorder different to Parkinson's disease
* Patients, who are post-ictus and/or traumatic brain injury (TBI)
* Patients, who are treated with antipsychotic drugs
* Obese persons (BMI > 27)
* Idiopathic normal pressure idrocephalus (INPI)
* Paget's disease
* Breast cancer
* Adenocarcinoma of the prostate
* Glucose-6-phosphate (GSD-I) deficiency
* Insuline-resistance-related disorders

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the recruited subjects will be either healthy people group or patients with a defined diagnosis of Parkinson (classification of Hoehn and Yahr).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Waldner, MD, Study Director — Privatklinik Villa Melitta; Sarah Dassati, BSc, Principal Investigator — Privatklinik Villa Melitta
Locations (1):
- Privatklinik Villa Melitta, Bolzano, Südtirol, Italy

REFERENCES:
- [Background] Bennett MD. The time and duration of meiosis. Philos Trans R Soc Lond B Biol Sci. 1977 Mar 21;277(955):201-26. doi: 10.1098/rstb.1977.0012. PMID 16285
- [Background] Patterson D, Carnright DV. Biochemical genetic analysis of pyrimidine biosynthesis in mammalian cells: I. Isolation of a mutant defective in the early steps of de novo pyrimidine synthesis. Somatic Cell Genet. 1977 Sep;3(5):483-95. doi: 10.1007/BF01539120. PMID 21463
- [Background] Arnesen K, Nordstoga K. Ocular encephalitozoonosis (nosematosis) in blue foxes. Polyarteritis nodosa and cataract. Acta Ophthalmol (Copenh). 1977 Aug;55(4):641-51. doi: 10.1111/j.1755-3768.1977.tb05662.x. PMID 19918
- [Background] Weidler DJ, Sieck GC. A study of ion binding in the hemolymph of Periplaneta americana. Comp Biochem Physiol A Comp Physiol. 1977;56(1A):11-4. doi: 10.1016/0300-9629(77)90433-9. No abstract available. PMID 11058
- [Background] Bergdahl B, Andersson KE. Stability in vitro of methylproscillaridin. Eur J Clin Pharmacol. 1977 Apr 20;11(4):267-71. doi: 10.1007/BF00607675. PMID 16755
- [Background] Kovatsis A, Kovatsi-Kotsaki V, Elezoglou B, Kounenis G. Physiological antagonism between PGE2, PGA1, PGF1-alpha and NADP, beta-NAD on isolated rabbit jejunum. Arzneimittelforschung. 1976;26(11):1997-9. PMID 14647
- [Result] Shankar GM, Walsh DM. Alzheimer's disease: synaptic dysfunction and Abeta. Mol Neurodegener. 2009 Nov 23;4:48. doi: 10.1186/1750-1326-4-48. PMID 19930651
- [Result] Dalmark M. Chloride in the human erythrocyte: distribution and transport between cellular and extracellular fluids and structural features of the cell membrane. Prog Biophys Mol Biol. 1976;31(2):145-64. No abstract available. PMID 10601
- [Result] Miller J, Wallace D, Grieco MH, Frenkel R, Larsen K. Double-blind trial of oral carbuterol in bronchial asthma. Ann Allergy. 1977 Jul;39(1):12-7. PMID 18957
- [Result] Fall RR. Stabilization of an acetyl-coenzyme A carboxylase complex from Pseudomonas citronellolis. Biochim Biophys Acta. 1976 Dec 20;450(3):475-80. doi: 10.1016/0005-2760(76)90022-9. PMID 12801
- [Result] Hong JS. An ecf mutation in Escherichia coli pleiotropically affecting energy coupling in active transport but not generation or maintenance of membrane potential. J Biol Chem. 1977 Dec 10;252(23):8582-8. No abstract available. PMID 21876
- [Result] Kricka LJ, Carter TJ. A method for enhancing the stability of thiol-containing enzymes immobilised on nylon. Clin Chim Acta. 1977 Aug 15;79(1):141-7. doi: 10.1016/0009-8981(77)90471-5. PMID 19176
- See also: Participating Centre for ApoD Detection — http://www.villamelitta.it

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 healthy subjects are enrolled on the base of their age being classified in the groups I (20-40), II (40-65) and three (>than 65). 90 patients are enrolled on the base of their disease's stage (Hoehn and Yahr classification) being classified in the groups A (I, H&Y), B (II, H&Y) and C (> than II, H&Y).
Groups:
- Group I: 30 Healthy Subjects aged 20-40
- Group II: 30 Healthy Subjects aged 40-65
- Group III: 30 Healthy Subjects aged more than 65
- Group A: 30 Patients at Stage I, H&Y classification
- Group B: 30 Patients at Stage II, H&Y classification
- Group C: 30 Patients at Stage more than III, H&Y classification
Period: Overall Study
Arm/Group | Group I | Group II | Group III | Group A | Group B | Group C
Started | 30 | 30 | 30 | 30 | 30 | 30
Completed | 30 | 30 | 30 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 30 | 30 | 30
Not completed — Enrollment of patients (PD) in 09/2013 | 0 | 0 | 0 | 30 | 30 | 30

BASELINE CHARACTERISTICS:
Groups:
- Group A: Patients at Stage I, H&Y
- Group B: Patients at Stage II, H&Y
- Group C: Patients at stage > than II, H&Y
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Group A | Group B | Group C | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30 | 30 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 0 | 0 | 0 | 0 | 60
  >=65 years | 0 | 0 | 30 | 30 | 30 | 30 | 120
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 15 | 15 | 15 | 90
  Male | 15 | 15 | 15 | 15 | 15 | 15 | 90
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 30 | 30 | 30 | 30 | 30 | 180

OUTCOME MEASURES:

1. Primary Outcome: Detection of Apolipoprotein D
Description: Apolipoprotein D (apoD)concentration in human serum as a potential marker for Parkinson's disease (PD)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: microg / ml
Arm/Group | Group I | Group II | Group III | Group A | Group B | Group C
Number analyzed (Participants) | 30 | 30 | 30 | 0 | 0 | 0
microg / ml | 28.28 (4.01) | 27.73 (7.26) | 34.61 (9.21) |  |  |

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events weren not collected/assessed
Arm/Group | Group I | Group II | Group III | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No